CLINICAL TRIAL: NCT03105037
Title: The Effect of Supraglottic Airway Insertion on the Accuracy of Cricothyroid Membrane Identification in Females- a Prospective Observational Study.
Brief Title: The Effect of Supraglottic Airway Insertion on the Accuracy of Cricothyroid Membrane Identification in Females
Status: Completed | Type: Observational
Sponsor: The Rotunda Hospital (Other)
Responsible Party: Principal Investigator, Tom Drew, Principal Study Investigor, SpR Anaesthetist, The Rotunda Hospital
Other Study IDs: REC-2017-001
Record Dates: First submitted 2017-03-25; First posted 2017-04-07 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Airway Obstruction
MeSH Terms: conditions — Airway Obstruction

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: CTM assessed with supraglottic airway in situ and without

SUMMARY:
Prospective, observational, study that will examine if a sited supraglottic airway (the igel) will increase the accuracy of identifying the cricothyroid membrane in female patients.

Consented patients that meet inclusion criteria are assessed by clinicians under general anaesthesia with and without a supraglottic airway in situ. The accuracy of CTM identification by palpation will be evaluated using ultrasound.

DETAILED DESCRIPTION:
Palpation of the airway structures results in misidentification of the cricothyroid membrane (CTM) in a high proportion of women. Female front of neck anatomy is less distinct compared to males with reduced angulation of the laryngeal cartilages making it harder to distinguish the relevant landmarks. In obese patients, overlying subcutaneous tissue compounds this problem and several studies have demonstrated poor success identifying the CTM by palpation in this population. Supraglottic airway device (SAD) insertion precedes emergency front of neck access attempts in the stepwise progression from failed intubation to cricothyroidotomy. The nature and clinical implication of SAD insertion on cricothyroidotomy remain unstudied.

Sixty four patients will undergo front of neck airway assessment by volunteer clinicians with and without a SAD in situ (control and SAD assessments, within-subjects design). The patients are fasting women presenting for routine gynaecological surgery. Eight anaesthetists, at different levels of training, will perform eight individual CTM assessments with and without the SAD in situ.

Ultrasound images will be captured in the sagittal plane immediately before and after supraglottic airway insertion. Images are then downloaded, anonymised and randomised for blinded digital analysis.

ELIGIBILITY:
Inclusion Criteria:

* Women attending for routine surgery

Exclusion Criteria:

* unable to give informed consent
* abnormal neck anatomy
* history of gastroesophageal reflux
* history of neck surgery or radiotherapy
* contraindication to supraglottic airway device insertion

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: women attending for routine gynaecological surgery
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2017-01-31 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
accurate identification of the cricothyroid membrane | At clinician assessment, on the day of patient recruitment.
  accuracy of cricothyroid membrane identification, measured as either successful identification or unsuccessful (binary outcome). A successful identification is within 5mm of the midline and within the upper and lower borders of the cricothyroid membrane as measured using ultrasound.

SECONDARY OUTCOMES:
Accurate identification of the midline of the neck | At clinician assessment, on the day of patient recruitment.
  Accurate identification of the midline of the neck, binary outcome. A successful identification is within 5mm of the midline of the cricothyroid membrane as measured using ultrasound.
Difficulty of cricothyroid membrane assessment | At clinician assessment, on the day of patient recruitment.
  Difficulty of assessing the cricothyroid membrane as graded subjectively by the clinician using a visual analogue scale (VAS) where '0' is the easiest possible assessment of the location of the cricothyroid membrane and '10' is the most difficult possible assessment of the location of the cricothyroid membrane.
Time taken to attempt localisation of the cricothyroid membrane | At clinician assessment, on the day of patient recruitment.
  The time taken in seconds to attempt localisation of the cricothyroid membrane
Distance from clinician assessment to actual cricothyroid membrane location | On blinded, retrospective ultrasound analysis of images captured at the time of clinician assessment of the cricothyroid membrane. Blinded retrospective ultrasound assessment is to take place within 3 months of patient recruitment
  The distance measured from the clinicians estimate of where the cricothyroid membrane is to where the actual location of the CTM is using ultrasound and measured in millimetres
The distance from the skin to the first tracheal ring | On blinded, retrospective ultrasound analysis of images captured at the time of clinician assessment of the cricothyroid membrane. Blinded retrospective ultrasound assessment is to take place within 3 months of patient recruitment
  The distance from the skin to the superficial surface of the first tracheal ring measured in millimetres using digital analysis of ultrasound images
The distance from the skin to the cricoid cartilage | On blinded, retrospective ultrasound analysis of images captured at the time of clinician assessment of the cricothyroid membrane. Blinded retrospective ultrasound assessment is to take place within 3 months of patient recruitment
  The distance from the skin to the superficial surface of the first tracheal ring measured in millimetres using digital analysis of ultrasound images
The angle between the surface tissue interface of the cricothyroid membrane and the trachea | On blinded, retrospective ultrasound analysis of images captured at the time of clinician assessment of the cricothyroid membrane. Blinded retrospective ultrasound assessment is to take place within 3 months of patient recruitment
  The angle between the surface tissue interface of the cricothyroid membrane and the trachea measured in degrees using digital analysis of ultrasound images

CONTACTS AND LOCATIONS:
Overall Officials: Conan McCaul, Study Director — Prof
Locations (1):
- The Rotunda Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No